CLINICAL TRIAL: NCT04087824
Title: Development and Validation of a Deep Learning Algorithm for Real-time Recognition of Colonic Segments.
Brief Title: Deep Learning Algorithm for Recognition of Colonic Segments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019SDU-QILU-G003
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Colonic Diseases
Keywords: Deep learning; Colonoscopy; Central Neural Networks
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI monitoring colonoscopy (Experimental): Patients in this group go through colonoscopy under the AI monitoring device.
  Interventions: Device: AI assisted recognition of colonic segments

INTERVENTIONS:
Device: AI assisted recognition of colonic segments — After receiving standard bowel preparation regimen, patients go through colonoscopy under the AI monitoring device. The whole withdrawal process is monitored by AI associated recognition system. Key colonic segments include ileocecal valve, ascending colon, transverse colon, descending colon, sigmoid colon and rectum. When typical anatomic sites are detected, the AI device will automatically captured relevant images and report the name of each segment on the screen. The operating endoscopy expert will give the final answer and judge the performance of AI, which is set as a golden standard. Then all the AI captured images will be reviewed by human group, which consists of three to five experienced endoscopic physicians.

SUMMARY:
The purpose of this study is to develop and validate a deep learning algorithm to realize automatic recognition of colonic segments under conventional colonoscopy. Then, evaluate the accuracy this new artificial intelligence(AI) assisted recognition system in clinic practice.

DETAILED DESCRIPTION:
Colonoscopy is recommended as a routine examination for colorectal cancer screening. Complete inspection of all colon segments is the basis of colonoscopy quality control, and furthermore improves the detection rates of small adenomas. Recently, deep learning algorithm based on central neural networks (CNN) has shown multiple potential in computer-aided detection and computer-aided diagnose of gastrointestinal lesions. However, there is still a blank in recognition of anatomic sites, which restricts the realization of AI-aided lesions detection and disease severity scoring. This study aim to train an algorithm to recognize key colonic segments, and testify the accuracy of each segments recognition as compared to endoscopic physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years undergoing conventional colonoscopy

Exclusion Criteria:

* Known or suspected bowel obstruction, stricture or perforation
* Compromised swallowing reflex or mental status
* Severe chronic renal failure(creatinine clearance < 30 ml/min)
* Severe congestive heart failure (New York Heart Association class III or IV)
* Uncontrolled hypertension (systolic blood pressure > 170 mm Hg, diastolic blood pressure > 100 mm Hg)
* Dehydration
* Disturbance of electrolytes
* Pregnancy or lactation
* Hemodynamically unstable
* Unable to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
The accuracy of each colonic segment real-time recognition with deep learning algorithm. | 3 months.
  The segmental recognition accuracy is the proportion of correctly recognized segments divided by the number of involved patients. The accuracy rate of ileocecal valve, ascending colon, transverse colon, descending colon, sigmoid colon and rectum will be separately calculated.

SECONDARY OUTCOMES:
The accuracy of total colonic segments recognition with deep learning algorithm as compared to endoscopic experts group. | 3 months.
  The total recognition accuracy is the proportion of correctly recognized images divided by the number of AI captured images. Then all AI captured images will be reviewed by experts group to give a human evaluating rate. Two rates will be compared by student t test to analyze the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University